CLINICAL TRIAL: NCT03145870
Title: Prevalence of Asymptomatic Thrombosis in Multiple Myeloma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2014_843_0009
Record Dates: First submitted 2017-05-04; First posted 2017-05-09 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Thrombosis; Multiple Myeloma
MeSH Terms: conditions — Thrombosis; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with multiple symptomatic myeloma (Other)
  Interventions: Other: Echoing of the lower limbs and measuring the systolic pressure index

INTERVENTIONS:
Other: Echoing of the lower limbs and measuring the systolic pressure index — Echoing of the lower limbs and measuring the systolic pressure index

SUMMARY:
Malignant hemopathies, such as solid cancers, increase the risk of venous and arterial thromboembolic events. The incidence of symptomatic venous thromboembolic events is particularly high in myeloma, linked to the usual risk factors for venous thromboembolic disease, biological risk factors specific to myeloma, and especially to its treatments.

The prevalence of asymptomatic venous thromboembolic events and arterial events are not known to date and remain important data for planning a possible randomized study to determine the most suitable thromboprophylaxis in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient major age ≥18 years
* Patients with symptomatic myeloma meeting the definition of the International Myeloma Working Group, regardless of the therapeutic line, including patients in remission and untreated.
* Patient having given informed consent, signed.
* Patient benefiting from a social security scheme

Exclusion Criteria:

* Patients with non-symptomatic myeloma (stage I) or gammapathy of unknown significance (MGUS).
* Patient undergoing antithrombotic treatment for deep or superficial venous thrombosis and / or pulmonary embolism at the time of inclusion.
* Patients with occlusive arterial disease of the lower limbs known at the time of inclusion.
* Minors, protected adults and patients deprived of liberty or not affiliated to a social security scheme
* Pregnant woman
* Patient unable to express consent.
* Patient under guardianship or curatorship or patient deprived of public liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Analysis of the occurrence of venous thromboembolic events via transverse Doppler echo | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France